CLINICAL TRIAL: NCT03077217
Title: Low-dose Rifaximin in the Treatment of Covert Hepatic Encephalopathy: A Randomized Open Controlled Study
Brief Title: Low-dose Rifaximin in the Treatment of Covert Hepatic Encephalopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Wei-Fen Xie, Director, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CZH0010
Record Dates: First submitted 2017-01-30; First posted 2017-03-10 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Covert Hepatic Encephalopathy
Keywords: covert hepatic encephalopathy; low-dose rifaximin
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- the high-dose rifaximin (Active Comparator): The high-dose rifaximin group was given rifaximin 1200 mg/day for 8 weeks.
  Interventions: Drug: Rifaximin
- the low-dose rifaximinl group (Active Comparator): The low-dose rifaximin group was given rifaximin 800 mg/day for 8 weeks.
  Interventions: Drug: Rifaximin
- the control group (Placebo Comparator): The control group didn't receive rifaximin treatment
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — The investigators use low-dose rifaximin for the treatment of patients with covert hepatic encephalopathy

SUMMARY:
Several studies have been showed that rifaximin can improve cognitive functions, driving simulator performance and health-related quality of life in patients with minimal hepatic encephalopathy. The aim of this prospective randomized open controlled study was to evaluate the efficacy and safety of rifaximin at different doses for the treatment of covert hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients agreed to sign the informed consents
2. Patients aged 18-70 years，males or females
3. Patients who were diagnosed with occult hepatic encephalopathy by PHES and Stroop tests

Exclusion Criteria:

1. Allergy to rifamycin/rifamutin/rifampin/rifapentine
2. Current or recent (<3 month) use of alcohol or can't stop drinking during the study period
3. Use of antibiotics within last 6 weeks
4. Use of lactulose/lactitol, probiotics, L-ornithine-L-aspart，zinc，metronidazole, neomycin, or rifaximin within last 6 weeks
5. Infection or gastrointestinal hemorrhage within last 6 weeks
6. Use of psychoactive drugs within last 6 weeks
7. Occurred overt hepatic encephalopathy within last 3 months
8. history of portosystemic shunt surgery or transjugular intrahepatic portosystemic shunt
9. Poor vision, color blindness or motor defects that interfere with the performance of psychometric tests
10. Other non-controllable neurological or psychiatric problems which may affect cognitive function such as Alzheimer's disease, Parkinson's disease or schizophrenia
11. Conformed or highly suspicious diagnosis of liver malignant tumors
12. Human immunodeficiency virus (HIV) infection
13. Uncontrolled hypertension, diabetes or other serious cardiac and pulmonary diseases
14. White blood cell count<1×10^9/L
15. Pregnancy and breastfeeding
16. Participated in other drug clinical trials within 3 months
17. The researchers thought it was not suitable for this clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients showing covert hepatic encephalopathy reversal | up to 6 months
  the percentage of patients showing covert hepatic encephalopathy reversal
health-related quality of life improvement | up to 6 month
  complete the questionnaire "sickness impact profile"

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180